CLINICAL TRIAL: NCT05634603
Title: Efficacy of Lactose-free Milk in Treating Acute Gastroenteritis in Infants: A Randomised Controlled Trial
Brief Title: Efficacy of Lactose-free Milk in Treating Acute Gastroenteritis in Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Women and Children Hospital of An Giang (Other)
Collaborators: Can Tho University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Rang Nguyen, University of Medicine and Pharmacy of Can Tho, The Women and Children Hospital of An Giang
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WCHAnGiang
Record Dates: First submitted 2022-11-21; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Acute Gastroenteritis
Keywords: diarrhea lactose-free diet

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Lactose-free milk formula (Frisolac LF ®)
  Interventions: Dietary Supplement: Lactose-free milk formula (Frisolac LF ®)
- Placebo (Placebo Comparator): Regular infant milk formula
  Interventions: Dietary Supplement: Lactose-free milk formula (Frisolac LF ®)

INTERVENTIONS:
Dietary Supplement: Lactose-free milk formula (Frisolac LF ®) — Following the initial rehydration phase, children were alternately assigned to receive 100 ml/kg/day of either lactose-free or lactose-containing formula

SUMMARY:
The purpose of this study is to determine whether lactose-free milk will change diarrhea duration and severity in formula-fed infants with acute gastroenteritis presenting to pediatric wards.

DETAILED DESCRIPTION:
More than 525 000 children die each year due to diarrheal disease, the second leading cause of death among children under five. Children from Asian countries, including Vietnamese children, frequently have lactose intolerance. In addition, gastroenteritis, specifically rotavirus-induced gastroenteritis, temporarily impairs lactase enzymes in the intestines. In a recent Cochrane review of 33 randomized and quasi-randomized trials, lactose-free diets reduced diarrhea among children younger than 5 years old. These trials, however, involved inpatients in middle-or high-income countries. Neither patient was from a developing country, where diarrheal diseases often cause significant morbidity and mortality. The purpose of this study is to determine whether lactose-free milk will change the duration and severity of diarrhea in Vietnamese infants with acute gastroenteritis.

ELIGIBILITY:
Inclusion Criteria:

* Children 2- 24 months old on artificial milk formula
* Acute diarrhea (3 or more loose or liquid stools per day)

Exclusion Criteria:

* Used antibiotics within 3 days before admission
* Breastfeeding
* Severe dehydration, defined by a need of IV rehydration
* Malnutrition (weight/height< -3SD)
* Chronic underlying disease, immunocompromised condition or systemic infection

Ages: 2 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in diarrhea duration | 7 days
  llness onset and last diarrhoeal stool (the number of days with 3 or more loose or watery stools)

SECONDARY OUTCOMES:
Weight gain | 7 days
Severity of diarrhea according to the modified Vesikari score | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Can Tho Children Hospital, Can Tho, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] MacGillivray S, Fahey T, McGuire W. Lactose avoidance for young children with acute diarrhoea. Cochrane Database Syst Rev. 2013 Oct 31;2013(10):CD005433. doi: 10.1002/14651858.CD005433.pub2. PMID 24173771
- [Result] Simakachorn N, Tongpenyai Y, Tongtan O, Varavithya W. Randomized, double-blind clinical trial of a lactose-free and a lactose-containing formula in dietary management of acute childhood diarrhea. J Med Assoc Thai. 2004 Jun;87(6):641-9. PMID 15279342